CLINICAL TRIAL: NCT03087981
Title: A Multicenter Prospective Observational Study to Analyze Various ICP Derived Parameters and Clinical Status in Neurosurgical Critical Patients Through Big Data Acquisition
Brief Title: Parameters Analysis in Neurosurgical Critical Patients Through Big Data Acquisition
Acronym: PANDA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Renjineuro-BDA(2017)
Record Dates: First submitted 2017-03-12; First posted 2017-03-23 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-03

CONDITIONS: Intracranial Pressure; Neurosurgery; Information Management

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The PANDA trial is a multicenter prospective observational study designed to analyze various ICP derived parameters and clinical status in neurosurgical critical patients through a new big data acquisition system.

DETAILED DESCRIPTION:
Nowadays, intracranial pressure (ICP) monitoring is widely used as a way to evaluate intracranial status in neurosurgery department especially in neurosurgical critical patients. Most of us focus only on the mean ICP value while ignoring other ICP derived parameters, such ICP waveform, AMP, RAP, PRx, IAAC and so on. However, it is reported that these parameters can reflect the status of intracerebral circulation, cerebrospinal compensatory reserve and brain compliance and can often be indicative of impending neurological deterioration and even outcome of patients. The PANDA trial is a multicenter prospective observational study designed to investigate the relationship between these ICP derived parameters and clinical status and to uncover the mechanism behind it. We will use a brand-new automatic big data collecting and storing system to continuously acquire patients' physiological information such as blood pressure, ICP, ETCO2，EEG etc. before analysis. Hopefully, this trial will reveal what is happening in the cranial cavity through the natural history of different kinds of intracranial lesion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old
* Intracranial lesion underwent ICP sensor implantation
* Informed consent obtained

Exclusion Criteria:

* No consent
* A life-threatening injury to an organ other than the brain
* Known pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with intracranial lesion
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Glasgow Outcome Scale(GOS) | within 3 months after enrollment
Glasgow Coma Scale(GCS) | within 3 months after enrollment
Disability Rating Scale (DRS) | within 3 months after enrollment
Mean intracranial pressure(ICP) value | throughout ICP monitoring, average 7 days
Correlation between pulse amplitude and mean intracranial pressure(RAP) | throughout ICP monitoring, average 7 days
Pressure-reactivity index(PRx) | throughout ICP monitoring, average 7 days
Pulse amplitude of ICP(AMP) | throughout ICP monitoring, average 7 days
ICP-arterial blood pressure(ABP) wave amplitude correlation(IAAC) | throughout ICP monitoring, average 7 days
Cerebral perfusion pressure(CPP) | throughout ICP monitoring, average 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Di Ieva A, Schmitz EM, Cusimano MD. Analysis of intracranial pressure: past, present, and future. Neuroscientist. 2013 Dec;19(6):592-603. doi: 10.1177/1073858412474845. Epub 2013 Feb 6. PMID 23389057
- [Background] Eide PK, Sorteberg A, Bentsen G, Marthinsen PB, Stubhaug A, Sorteberg W. Pressure-derived versus pressure wave amplitude-derived indices of cerebrovascular pressure reactivity in relation to early clinical state and 12-month outcome following aneurysmal subarachnoid hemorrhage. J Neurosurg. 2012 May;116(5):961-71. doi: 10.3171/2012.1.JNS111313. Epub 2012 Feb 10. PMID 22324419
- [Background] Czosnyka M, Smielewski P, Timofeev I, Lavinio A, Guazzo E, Hutchinson P, Pickard JD. Intracranial pressure: more than a number. Neurosurg Focus. 2007 May 15;22(5):E10. doi: 10.3171/foc.2007.22.5.11. PMID 17613228
- [Background] Czosnyka M, Pickard JD. Monitoring and interpretation of intracranial pressure. J Neurol Neurosurg Psychiatry. 2004 Jun;75(6):813-21. doi: 10.1136/jnnp.2003.033126. PMID 15145991
- [Background] Hamilton R, Xu P, Asgari S, Kasprowicz M, Vespa P, Bergsneider M, Hu X. Forecasting intracranial pressure elevation using pulse waveform morphology. Annu Int Conf IEEE Eng Med Biol Soc. 2009;2009:4331-4. doi: 10.1109/IEMBS.2009.5332749. PMID 19963821